CLINICAL TRIAL: NCT02030548
Title: Bleeding in Patients Undergoing Urgent CABG During Dual Antiplatelet Therapy Including the New P2Y12 Receptor Inhibitors Prasugrel and Ticagrelor
Brief Title: Bleeding in Patients Undergoing CABG (Coronary Artery Bypass Graft) During Dual Antiplatelet Therapy
Status: Terminated | Type: Observational
Why Stopped: enrolment behind expectation
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: NIS003684
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Acute Coronary Syndrome
Keywords: CABG; dual antiplatelet therapy; aspirin; clopidogrel; prasugrel; ticagrelor
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute CABG: patients undergoing acute CABG with or without valve replacement during dual antiplatelet therapy

SUMMARY:
The aim of the study is to evaluate surgery-related bleeding and mortality in patients needing acute coronary artery bypass grafting with or without valve replacement during dual antiplatelet therapy with aspirin and a P2Y12 receptor blocker (Clopidogrel, Prasugrel, Ticagrelor)

ELIGIBILITY:
Inclusion Criteria:

consecutive patients undergoing acute CABG with or without valve replacement within 7 days after last intake of dual antiplatelet therapy

Exclusion Criteria:

concomitant oral anticoagulants dialysis surgery employing hypothermic cardiac arrest

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing acute CABG with or without valve during dual antiplatelet therapy
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
calculated blood loss | until postoperative day 5

SECONDARY OUTCOMES:
mortality | from index surgery until one year after index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Mahla, MD, Principal Investigator — Dept. of Anesthesiology and Intensive Care Medicine, MUG
Locations (1):
- Dept. of Anesthesiology and Intensive Care Medicine, Graz, Styria, Austria